CLINICAL TRIAL: NCT04149522
Title: Mepitel Film® Prophylaxis For Breast Cancer Patients Receiving Breast Radiotherapy At High Risk For Moist Desquamation: A Phase II Study
Brief Title: Evaluation of Mepitel Film® in Preventing Epidermitis in Patients Receiving Radiation Therapy for Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The mepitel film was expired and was no longer available.
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Principal Investigator, Mark Trombetta, MD, MD, Radiation Oncology, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-185-AGH
Record Dates: First submitted 2019-10-22; First posted 2019-11-04 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer; Radiotherapy; Adverse Effect, Dermatitis or Eczema; Radiotherapy Side Effect; Radiation Burn; Radiation Dermatitis; Radiotherapy; Complications
Keywords: Radiotherapy breast; Mepitel Film
MeSH Terms: conditions — Breast Neoplasms; Dermatitis; Eczema; Radiation Injuries; Radiodermatitis

STUDY DESIGN:
Intervention Model Description: 2 study arms - 20 women to receive Mepitel film on medial aspect of breast, 20 women to receive Mepitel film on lateral aspect of breast
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Medial Breast Tissue (Active Comparator): Women assigned to the medial breast tissue arm, will have the area of the breast visually divided into 2 equal parts; medial and lateral. The film will be applied to the medial breast tissue by clinically trained staff on day 1 of radiotherapy, the lateral segment will not be covered. The treatment area is cleaned with mild soap, rinsed with water, and dried. The film is applied, sticky side to the skin, then the paper frame is removed. Multiple sheets of non-overlapping film will be used to adequately cover the treatment area. During course of radiotherapy, new film may be applied by clinically trained staff in the event the film no longer adheres to the skin or comes off. Replacement of the film may be done as often as necessary. If there are signs of infection (e.g. redness, feeling warm or swollen), film can be removed. The film will remain in place until one week following the last day of radiotherapy, where it will be removed by the physician or clinically trained staff.
  Interventions: Device: Mepitel Film®
- Lateral Breast Tissue (Active Comparator): Women assigned to the lateral breast tissue arm will have the area of the breast visually divided into 2 equal parts; medial and lateral. The film will be applied to the lateral breast tissue only, by trained staff on day 1 of radiotherapy. The in-field ipsilateral axilla will be included with lateral breast segment to extent necessary to cover breast or chest wall only. The skin is cleaned with mild soap, rinsed with water, and dried. The film is applied, sticky side to skin and paper frame is removed. Multiple sheets of non-overlapping film will be used to cover the treatment area. During course of therapy, new film may be applied as often as necessary, by trained staff if film no longer adheres to skin or comes off. If there are signs of infection (e.g. redness, feeling warm or swollen), the film can be removed. The film will remain in place until one week following the last day of radiotherapy, where it will be removed by the physician or trained staff.
  Interventions: Device: Mepitel Film®

INTERVENTIONS:
Device: Mepitel Film® — As a part of this research study, Mepitel Film® will be placed prior to a participant's first radiation treatment, and will be removed one week following the end of treatment. The Film will be placed by the physician or his/her designee to cover approximately one-half of the breast divided in the cephalo-caudal plane. The film will remain in place until one week following the completion of radiotherapy. Any loss of film applied will be replaced as needed. Application of the Film is done by research personnel clinically trained in its application procedures.

SUMMARY:
The purpose of this research is to evaluate the use of Mepitel Film® in preventing radiation epidermitis in patients receiving radiation treatment for breast cancer. Mepitel® Film is a thin, flexible, waterproof, and breathable film made of a soft silicone layer and polyurethane film. Mepitel ® film is not made with natural rubber latex (NRL). It is FDA approved for the management of superficial wounds, such as superficial burns. As a part of this research study, the Mepitel Film® will be placed prior to participant's first radiation treatment, and will be removed one week following the end of treatment. Throughout the study, information will be collected to analyze at the end of the research study to determine if the Mepitel Film® helps prevent skin breakdown. The subjects will be followed per standard of care and examined for skin redness, warmth or swelling as normally examined and cared for during standard radiation therapy. If radiation burns are noted, the subject will be treated normally and depending on the severity of the radiation burns, may be removed from the study treatment and treated through standard of care.

DETAILED DESCRIPTION:
Clinical Phase II trial to determine if Mepitel Film® is a viable prophylactic option for high-risk women undergoing radiotherapy for breast cancer to reduce side effects of radiation on the skin.

The objective of this study is to evaluate the efficacy of use of Mepitel Film® in the prevention of grade II or higher radiation epidermitis in high-risk patients undergoing radiotherapy for breast cancer.

Test Article(s) Mepitel Film ®

The proposed study is a cohort trial of women with breast cancer who are at a high risk of having pain, swelling, inflammation with skin tenderness, skin ulceration, pruritis, and scarring during radiation treatment.

Each subject's participation will last approximately eight weeks. The entire study is expected to last up to 24 months.

The primary analysis will be based classification of radiation dermatitis from treated and untreated skin at each visit. Secondary endpoints will review quality of life responses compared to dermatitis.

Statistical analysis will be completed by Highmark Health Data Science R&D. The principal investigator will share any updates, AEs and safety concerns to the Data Safety Monitoring Board (DSMB), a group of scientists, physicians, statisticians, and others that collect and analyze data during the course of a research study to monitor for adverse events and other trends that would warrant modification or termination of the trial or notification of subjects about new information that might affect their willingness to continue in the trial. The Highmark Health Data Science Research and Development department are the statisticians for this study and will participate on the DSMB.

General Schema of Study Design Women who meet inclusion/exclusion for the trial and are consent to participate in the trial are enrolled in the study. Prior to standard of care radiation treatments, women will have the area of the breast divided into two, approximately equal parts; medial and lateral. The in-field ipsilateral axilla will be included with the lateral breast segment to the extent necessary for coverage of the breast or chest wall only. The infra-mammary crease will be part of both the medial and lateral breast segments. Axillary irradiation is allowed and the nodal areas irradiated should be considered as part of the evaluable field and covered with the Film as required by division of the breast as above. The aspect of the breast covered by the Mepitel Film® will alternate with consecutive patients and the axilla will be separately evaluated for acute reaction. Each woman will act as her own control. The breast will be photographed (digital images). At each treatment, the breast will be evaluated for signs of infection, erythema, induration, dry or wet desquamation or frank skin breakdown. A Quality-Of-Life (QOL) Instrument will be completed by the patient.

All radiotherapy visits are standard of care for participants. The Mepitel Film® has been purchased for this study by the Allegheny General Hospital (AGH) Auxiliary and each box of Film received will be then labeled for investigational use only.

Study Duration, Enrollment and Number of Sites Length of time on study is dependent upon the radiotherapy regimen (25 fractions or 28 fractions) and any AE probably or definitely related to study participation. The expected length of time on study is 6 - 7 weeks: 25 to 28 business days (Monday-Friday) for the radiotherapy plus the one week post treatment follow up visit. Visits related to an adverse event (AE) will continue until the AE is resolved, which may extend participation time.

The study will be conducted at approximately 5 investigative sites in the Allegheny Health Network and the accrual goal is 40 women.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 - 80 years of age
2. Biopsy-proven diagnosis of breast cancer (Stage 0 - II) with the breast tumor completely removed
3. Whole breast or chest wall irradiation with or without ipsilateral axillary radiotherapy
4. Women of child-bearing potential must use an effective form of birth control

Exclusion Criteria:

1. Women who are pregnant or lactating
2. Women with evident skin irritation or skin infection (i.e. active rash, pre-existing dermatitis) or known allergy to adhesives or tapes; or known allergy to the Mepitel Film®
3. Women with a chest abnormality that would preclude application of the Film;
4. Women who in the investigator's opinion are not capable of completing the trial or following trial procedures

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of use of Mepitel Film® in the prevention of grade II or higher radiation epidermitis in high-risk patients undergoing radiotherapy for breast cancer | 7 weeks from initiation
  The breast will be photographed and assessed at the beginning of therapy and at weeks 3, 5 and 6 the 3 (which will occur if clinically indicated) and one week following the completion of therapy. At each treatment, the breast will be evaluated by a physician for signs of infection, erythema, induration, dry or wet desquamation or frank skin breakdown, utilizing a Radiation Dermitis scale (NCI CTCAE v4.03) at each visit. The scale ranges from 0 to 4, with 0-being no change, 1-faint erythema or dry desquamation, 2-moderate to brisk erythema, 3-confluent moist desquamation, 4-skin necrosis or ulceration, as assessed by the physician. The primary analysis will be based on the classification of radiation dermatitis from treated and untreated skin at each visit and will be analyzed using a chi-square or Fisher's Exact test as appropriate. Analysis will be stratified by any significant confounding factors or effect modifiers.

SECONDARY OUTCOMES:
Quality of Life (QOL) responses | 7 weeks from initiation
  A QOL questionnaire will be completed by each patient prior to first radiation treatment and at weeks 3, 5 and 6 (which will occur if clinically indicated) of radiotherapy, and 1 week following the completion of irradiation. The questionnaire asks subjects to rate symptoms on a scale from 1 to 4 (1 being excellent or no side effect to 4 being poor or worst side effect). The symptoms include: nipple appearance, arm movement, breast tenderness, breast swelling, breast sensitivity, swelling of breast, breast warm to touch, breast skin is red, breast skin is tanned, breast skin is flaking or peeling, breast itching, blisters or breast skin moist and raw, sharp shooting pains in the breast. Subjects will also be asked to choose the word (with definition) that best describes how their breast looks (excellent, good, poor or fair). Data will be analyzed using McNemar's test to compare the pre/post differences in survey response. Analysis will be stratified by any significant confounders.
Time until the onset of erythema | 7 weeks from initiation
  Time until onset of erythema with and without the film will be measured in days, based upon physician's physical exam and assessments at baseline and at each follow up visit. The breast will be photographed and assessed at the beginning of therapy and at weeks 3, 5 and 6 the 3 (which will occur if clinically indicated) and one week following the completion of therapy. At each treatment, the breast will be evaluated by a physician for signs of infection, erythema, induration, dry or wet desquamation or frank skin breakdown, utilizing a Radiation Dermitis scale (NCI CTCAE v4.03) at each visit. The scale ranges from 0 to 4, with 0-being no change, 1-faint erythema or dry desquamation, 2-moderate to brisk erythema, 3-confluent moist desquamation, 4-skin necrosis or ulceration, as assessed by the physician.
Time to healing skin treated with and without the film | 7 weeks from initiation
  Time to healing skin treated with and without the film will be measured in days, based upon physician's physical exam and assessments at baseline and at each follow up visit. The breast will be photographed and assessed at the beginning of therapy and at weeks 3, 5 and 6 the 3 (which will occur if clinically indicated) and one week following the completion of therapy. At each treatment, the breast will be evaluated by a physician for signs of infection, erythema, induration, dry or wet desquamation or frank skin breakdown, utilizing a Radiation Dermitis scale (NCI CTCAE v4.03) at each visit. The scale ranges from 0 to 4, with 0-being no change, 1-faint erythema or dry desquamation, 2-moderate to brisk erythema, 3-confluent moist desquamation, 4-skin necrosis or ulceration, as assessed by the physician.
Reduction in erythema | 7 weeks from initiation
  Reduction in erythema will be measured in percent change, based upon physician's physical exam and assessments at baseline and at each follow up visit. The breast will be photographed and assessed at the beginning of therapy and at weeks 3, 5 and 6 the 3 (which will occur if clinically indicated) and one week following the completion of therapy. At each treatment, the breast will be evaluated by a physician for signs of infection, erythema, induration, dry or wet desquamation or frank skin breakdown, utilizing a Radiation Dermitis scale (NCI CTCAE v4.03) at each visit. The scale ranges from 0 to 4, with 0-being no change, 1-faint erythema or dry desquamation, 2-moderate to brisk erythema, 3-confluent moist desquamation, 4-skin necrosis or ulceration, as assessed by the physician.
Reduction in moist desquamation | 7 weeks from initiation
  Reduction in moist desquamation will be measured in percent change, based upon physician's physical exam and assessments at baseline and at each follow up visit. The breast will be photographed and assessed at the beginning of therapy and at weeks 3, 5 and 6 the 3 (which will occur if clinically indicated) and one week following the completion of therapy. At each treatment, the breast will be evaluated by a physician for signs of infection, erythema, induration, dry or wet desquamation or frank skin breakdown, utilizing a Radiation Dermitis scale (NCI CTCAE v4.03) at each visit. The scale ranges from 0 to 4, with 0-being no change, 1-faint erythema or dry desquamation, 2-moderate to brisk erythema, 3-confluent moist desquamation, 4-skin necrosis or ulceration, as assessed by the physician.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Trombetta, MD, Principal Investigator — AHN Research Institute
Locations (5):
- United States (5):
  - AHN Cancer Institute at Jefferson Hospital, Clairton, Pennsylvania
  - AHN Cancer Institute Forbes, Monroeville, Pennsylvania
  - AHN Allegheny General Hospital, Pittsburgh, Pennsylvania
  - AHN West Penn Hospital, Pittsburgh, Pennsylvania
  - AHN Wexford Health + Wellness Pavilion, Wexford, Pennsylvania

REFERENCES:
- [Background] Herst PM, Bennett NC, Sutherland AE, Peszynski RI, Paterson DB, Jasperse ML. Prophylactic use of Mepitel Film prevents radiation-induced moist desquamation in an intra-patient randomised controlled clinical trial of 78 breast cancer patients. Radiother Oncol. 2014 Jan;110(1):137-43. doi: 10.1016/j.radonc.2014.01.005. Epub 2014 Jan 30. PMID 24486117